CLINICAL TRIAL: NCT07097207
Title: Study on the Efficacy and Safety of Autocrine p40 Chimeric Antigen Receptor T Cells Targeting CD19 and CD20 (CD19CD20-CAR.p40-T) in Refractory B-Cell Lymphoma
Brief Title: Efficacy and Safety of CD19CD20-CAR.p40-T in B-cell Lymphoma
Acronym: CAR-T
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 111; 111 (Other: Shenzhen Universisty general hospital)
Record Dates: First submitted 2025-07-11; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Relapsed/Refractory B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART group (Experimental): Participants will receive lymphodepleting chemotherapy (FC regimen: Fludarabine + Cyclophosphamide) on Days -5, -4, and -3 relative to the planned CD19/CD20-CAR.p40-T or CD19-CAR.p40-T cell infusion. The CAR-T cell infusion will be administered 72 hours after the completion of the FC chemotherapy.
  Interventions: Combination Product: CAR-T cell

INTERVENTIONS:
Combination Product: CAR-T cell — Participants will receive lymphodepleting chemotherapy (FC regimen: Fludarabine + Cyclophosphamide) on Days -5, -4, and -3 relative to the planned CD19/CD20-CAR.p40-T or CD19-CAR.p40-T cell infusion. The CAR-T cell infusion will be administered 72 hours after the completion of the FC chemotherapy.

SUMMARY:
1. Study Title:

   A Study on the Efficacy and Safety of Autocrine p40 CD19/CD20 Dual-Targeting Chimeric Antigen Receptor T-Cells (CD19/CD20-CAR.p40-T) in Relapsed/Refractory B-Cell Lymphoma
2. Study Objectives:

   * Primary Objective: To evaluate the safety of CD19/CD20 dual-targeting CAR.p40-T cell therapy in patients with relapsed/refractory B-cell lymphoma.
   * Secondary Objective: To evaluate the efficacy of CD19/CD20 dual-targeting CAR.p40-T cell therapy in patients with relapsed/refractory B-cell lymphoma.
3. Participant Intervention:

   * Participants will receive lymphodepleting chemotherapy (FC regimen: Fludarabine + Cyclophosphamide) on Days -5, -4, and -3 relative to the planned CD19/CD20-CAR.p40-T cell infusion or CD19 CAR.p40-T cell infusion. The CAR-T cell infusion will be administered 72 hours after the completion of the FC chemotherapy.

DETAILED DESCRIPTION:
A prospective, interventional Phase I/IIa clinical study to evaluate the safety and efficacy of autocrine p40 CAR-T cells targeting dual CD19/CD20 in refractory/relapsed B-cell lymphoma. A total of 20 patients aged 18 to 75 years with pathologically confirmed B-cell lymphoma (refractory/relapsed) will be enrolled. The total dose of CAR-T cells is 0.5-2×10^6 CAR-T cells/kg, administered as a single intravenous infusion. Eligible subjects (n=20) will be assigned by the investigator to receive either CD19CD20 CAR.p40-T injection or CD19 CAR.p40-T injection.

* Primary Endpoint**: To assess treatment-emergent adverse events (TEAEs) within 30 days after intravenous infusion of CAR-T cells.
* Secondary Endpoints**:

  * Objective response rate (ORR=CR+PR) within 8 weeks;
  * Overall survival (OS) and progression-free survival (PFS) at 6 months;
  * In vivo expansion and persistence kinetics of CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 15 and 75 years old, regardless of gender;
2. Diagnosed with relapsed/refractory B-cell lymphoma according to the 2020 World Health Organization (WHO) diagnostic criteria;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
4. Expected survival time of ≥ 3 months;
5. Confirmation of CD20 expression in tumor cells by flow cytometry/immunohistochemistry;
6. Patients tolerant to CD19 CAR-T cell therapy or those with low CD19 expression;
7. No severe heart, lung, liver, or kidney diseases;
8. Capable of understanding and willing to sign the informed consent form for this trial;
9. No contraindications to peripheral blood apheresis for the subject;
10. Having clearly measurable and evaluable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 standard;
11. The subject must have received standard first- and second-line treatment regimens;
12. Not having received antibody-based drug treatment within 2 weeks before cell therapy.

Exclusion Criteria:

1. History of allergy to any component in the cell product;
2. The following conditions in the blood routine examination: White blood cell count (WBC) ≤ 1×10⁹/L, absolute neutrophil count (ANC) ≤ 0.5×10⁹/L, absolute lymphocyte count (ALC) ≤ 0.5×10⁹/L, platelet count (PLT) ≤ 25×10⁹/L;
3. The following conditions in laboratory tests: including but not limited to, total serum bilirubin ≥ 1.5 mg/dl; serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the upper limit of normal; serum creatinine ≥ 2.0 mg/dl;
4. Patients with heart failure classified as grade III or IV according to the New York Heart Association (NYHA) classification criteria; or left ventricular ejection fraction (LVEF) < 50% as detected by echocardiography;
5. Abnormal lung function with oxygen saturation < 92% under room air;
6. Myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other clinically severe heart diseases within 12 months before enrollment;
7. Grade 3 hypertension with poorly controlled blood pressure despite drug treatment;
8. History of craniocerebral trauma, disturbance of consciousness, epilepsy, severe cerebral ischemia or intracerebral hemorrhagic diseases;
9. Patients with autoimmune diseases, immunodeficiency, or other conditions requiring immunosuppressive agent treatment;
10. Presence of uncontrolled active infection;
11. Previous use of any CAR-T cell product or other genetically modified T cell therapies;
12. Vaccination with live vaccines within 4 weeks before enrollment;
13. Subjects positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), and Treponema pallidum particle agglutination assay (TPPA)/rapid plasma reagin (RPR), as well as HBV carriers;
14. History of alcohol abuse, drug abuse, or mental illness in the subject;
15. The subject participated in any other clinical study within 3 months before joining this clinical study;
16. Female subjects with any of the following conditions: a) Currently pregnant or breastfeeding; or b) Having a pregnancy plan during the trial period; or c) Being fertile but unable to take effective contraceptive measures;
17. Other circumstances that, in the opinion of the investigator, make the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
TEAEs | From date of initial treatment to the 30 days after treatment
  Adverse events during treatment

SECONDARY OUTCOMES:
Disease-related clinical responses | From date of enrollment until the date of clinical responses,up to 2 years
  Disease-related clinical responses include CR/PR/SD/PD

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Wang, PHD, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Shenzhen University General Hospital, Shenzhen, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No